CLINICAL TRIAL: NCT06091202
Title: Tele-Collaborative Outreach to Rural Patients With Chronic Pain: The CORPs Trial
Brief Title: Tele-Collaborative Outreach to Rural Patients With Chronic Pain
Acronym: CORPs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Portland VA Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); North Texas Veterans Healthcare System (U.S. Federal Agency); VA Tennessee Valley Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Travis Lovejoy, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25384; 1UG3AT012257-01 (NIH); 4UH3AT012257-02 (NIH)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: Rural; Pain; CIH; Veteran
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CORPs Intervention (Active Comparator): The CORPs Intervention is a nurse-led intervention.
  A) An intake assessment with a Nurse Care Manager at the start of the study by phone or video to discuss the patient's pain experience, care options, and goals. Resources are provided and focus on non-medication options at the VA, and as appropriate, in the community.
  B) 5 Check-in phone/video appointments with a Nurse Care Manager, scheduled to take place near 2-, 4-, 8-, 12-, and 16-weeks. These visits will provide further assistance with goal planning and care coordination for pain management.
  C) Optional 6-week virtual group education class covering topics like complementary and integrative approaches to pain, sleep and pain, and the neurobiology of pain.
  D) Patients in this arm can contact their nurse with questions for the full 12 months of participation.
  Interventions: Behavioral: CORPs Intervention
- Minimally Enhanced Usual Care (MEUC) (Placebo Comparator): The minimally enhanced usual care arm is a one-time education session.
  A) One-time education session with a Nurse Care Manager by phone/video to review pain resources. These resources focus on non-medication options at the VA, and as appropriate, in the community.
  Interventions: Behavioral: Minimally Enhanced Usual Care (MEUC)

INTERVENTIONS:
Behavioral: CORPs Intervention — Participants will be randomly assigned to the intervention or to the comparator arm. The follow-up period is 12 months. The primary outcome is a change in pain interference.
  After the baseline assessment, participants will complete a masked telephone assessments with research staff at 3-, 6-, 9-, and 12-months.
  A subset of individuals may be invited to participate in a qualitative interview at 12-month follow-up.
  Other Names: Nurse-led collaborative care
  Arms: CORPs Intervention
Behavioral: Minimally Enhanced Usual Care (MEUC) — Participants will be randomly assigned to the intervention or to the comparator arm. The follow-up period is 12 months. The primary outcome is a change in pain interference.
  After the baseline assessment, participants will complete a masked telephone assessments with research staff at 3-, 6-, 9-, and 12-months.
  A subset of individuals may be invited to participate in a qualitative interview at 12-month follow-up.
  Other Names: One-time Education Session
  Arms: Minimally Enhanced Usual Care (MEUC)

SUMMARY:
This is a randomized controlled trial comparing the effectiveness of a remotely delivered collaborative care intervention for chronic pain versus a minimally enhanced control group. The specific aims of the study are: (1) compare the effectiveness of tele-collaborative pain care vs. minimally enhanced usual care to improve pain interference over 12 months of follow-up, and (2) oversample women and rural veterans of minoritized race/ethnicity to test heterogeneity of treatment effects across birth sex and race/ethnicity.

DETAILED DESCRIPTION:
The CORPs trial is a multisite pragmatic effectiveness trial taking place at four geographically diverse VA sites. The CORPs trial will assess the effectiveness of a nurse-led tele-collaborative pain care intervention (CORPs) compared to a one-time education session with a nurse (minimally enhanced usual care, or MEUC) at improving pain and health outcomes for Veterans living in rural areas. This study focuses on management of pain with non-medication services and therapies.

Veterans who enroll will participate for 12-months and will be randomized to one of 2 groups: 1) CORPs (with access to a nurse by phone/video for the duration of the study), or 2) One-time education session with the nurse by phone/video to review resources for pain. All participants complete research assessments at the start of the study, and at 3-, 6-, 9-, and 12-months by phone.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran
* Rural Residence based on Rural Urban Commuting Area codes
* High Impact Chronic pain, determined through a phone screening
* Access to landline or cell phone
* English Speaking

Exclusion Criteria:

* Cognitive impairment that would impact participation in the study
* Plans to move in the next 3 months
* Surgery in the past 3 months
* In long-term inpatient or hospice care
* Terminal illness (defined as life expectancy of less than 12 months)
* Active participation in another pain intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Interference - Brief Pain Inventory (BPI) | Baseline, 3-, 6-, 9-, and 12 Months
  Pain Interference subscale from the Brief Pain Inventory. Scores are reported on a range of 0 - 10, with higher scores indicating more impairment due to pain.

SECONDARY OUTCOMES:
Pain Intensity - Brief Pain Inventory (BPI) | Baseline, 3-, 6-, 9-, and 12 Months
  Scores are on a range of 0 - 10, with higher scores indicating more severe pain.
Physical Functioning - PROMIS Physical Functioning Scale | Baseline, 3-, 6-, 9-, and 12 Months
  Physical Functioning will be assessed with the 4-item PROMIS Physical Functioning scale. The physical function form asks the participant to rate a series of physical function related questions on a scale of 1-5 with one representing a better outcome.
Quality of Life - Veterans RAND-12 (VR-12) | Baseline, 3-, 6-, 9-, and 12 Months
  Quality of Life will be assessed with the Veterans RAND 12-item Health Survey (VR-12). VR-12 scores are summarized into two scores, a Physical Health component score and a Mental Health component score. Each component score is on a range of 0 - 100, with higher scores indicating more impairment in physical or mental health, respectively.
Depressive Symptoms - Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3-, 6-, 9-, and 12 Months
  Depressive symptoms will be assessed with the Patient Health Questionnaire-9 (PHQ-9). Scores on the PHQ-9 range from 0 - 24, with higher scores indicating more severe symptoms of depression.
Anxiety Symptoms - Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 3-, 6-, 9-, and 12 Months
  Anxiety symptoms will be assessed with the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Scores on the PHQ-9 range from 0 - 24, with higher scores indicating more severe symptoms of depression. Scores on the GAD-7 range from 0 - 21, with higher scores indicating more severe symptoms of anxiety.
Suicidal Behavior - Electronic Health Record (EHR) | Baseline, 3-, 6-, 9-, and 12 Months
  Data on suicidal behaviors will be extracted from the electronic health record.
Quality of Sleep - PROMIS Sleep Disturbance Scale | Baseline, 3-, 6-, 9-, and 12 Months
  Quality of sleep will be assessed with the PROMIS Sleep Disturbance 4-item short-form. The sleep disturbance form asks the participant to rate a series of sleep related questions on a scale of 1-5 with one representing a better outcome.
Engagement in Non-Pharmacological Services/Treatments - Nonpharmacological Self-Care Approaches survey (NSCAP) | Baseline, 3-, 6-, 9-, and 12 Months
  Engagement in nonpharmacological pain treatment will be assess with the Use of Nonpharmacological Self-Care Approaches survey (NSCAP). This survey assesses the number of times each of 9 treatments were used in the past 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Travis Lovejoy, PhD, MPH, Principal Investigator — Oregon Health & Science University, VA Portland Health Care System; Benjamin Morasco, PhD, Principal Investigator — Oregon Health & Science University, VA Portland Health Care System
Locations (4):
- United States (4):
  - VA Minneapolis Health Care System, Minneapolis, Minnesota
  - VA Portland Health Care System, Portland, Oregon
  - VA Tennessee Valley Health Care System, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No